CLINICAL TRIAL: NCT06588816
Title: The Correlation Between Pupil Size and Retinal Nerve Fibers Changes in Pseudoexfoliation Syndrome.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nayera Waleed Aboelwafa Mohamed, Resident, Assiut University
Other Study IDs: changes in pseudoexfoliation
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pseudoexfoliation Syndrome
Keywords: pupil; pseudoexfoliation; pupil dilation; pupil size; pseudoexfoliation syndrome
MeSH Terms: conditions — Exfoliation Syndrome; Mydriasis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: optical coherence tomography — Optical coherence tomography (OCT) is a non-invasive imaging test . It uses light waves to take cross-section pictures of the retina .
  With OCT, the ophthalmologist can see each of the retina's distinctive layers, and so we can use it to study the changes in pseudoexfoliation syndrome.

SUMMARY:
To study the possible correlation between pupillary diameter before and after dilation with intraocular pressure, lens stability and glaucomatous damage (represented by optic disc changes using cup to disc ratio and OCT changes in retinal nerve fiber layer and ganglion cell complex) in each eye of the same patient with PEX.

DETAILED DESCRIPTION:
Pseudoexfoliation (PEX) is a widespread condition that is often considered as a generalized disorder involving ocular manifestations as well as other body systems. It is characterized by the deposition of a distinctive fibrillar material in the anterior segment of the eye. The effect of pseudoexfoliation on various ocular tissues has been well studied in the past decades, especially both lens and optic disc damage. Key signs in pseudoexfoliative eyes are attributed to the effect of pseudoexfoliation material on pupillary muscles, lens and optic disc. Pseudoexfoliation appears to be a common disorder in older individuals in Upper Egypt with a prevalence of 4.14%. PXF was bilateral in 82.2% of cases. It was significantly associated with cataract, glaucoma and hearing loss. Of the PXF patients, 65% had cataract, 30.3% had glaucoma and 8.1% had hearing loss. Cardiovascular and cerebrovascular diseases such as angina, aortic aneurysm, and dementia have been linked to PXS. Subjects with PXF had a two- to three-fold increased risk for glaucoma according to the Blue Mountains Eye Study. The classic sign of PXF is the visualization of white pseudoexfoliative material on the pupil margin and on the anterior lens surface. It is believed that pupil size is another indicator for the severity of the disease. In this study we correlate the pupil size with other common ocular signs in PEX such as; lens subluxation and glaucomatous damage.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pseudoexfoliation syndrome.

Exclusion Criteria:

* previous ocular surgery or ocular trauma affecting the pupil. Any systemic or neurologic disease affecting the pupil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with pseudoexfoliation syndrome
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To study the possible correlation between pupillary diameter before and after dilation with intraocular pressure, lens stability and glaucomatous damage | Baseline
  in each eye of the same patient with PEX we study the correlation between the pupillary size before and after dilation with intraocular pressure, lens stability and glaucomatous damage represented by optic disc changes (cup to disc ratio) and OCT changes (RNFL and GCC).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tekin K, Kiziltoprak H, Sekeroglu MA, Yetkin E, Bayraktar S, Yilmazbas P. Static and dynamic pupil characteristics in pseudoexfoliation syndrome and glaucoma. Clin Exp Optom. 2020 May;103(3):332-338. doi: 10.1111/cxo.12945. Epub 2019 Jul 30. PMID 31364197
- [Background] Tuteja S, Zeppieri M, Chawla H. Pseudoexfoliation Syndrome and Glaucoma. 2023 May 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK574522/ PMID 34662036
- [Background] Katsi V, Pavlidis AN, Kallistratos MS, Fitsios A, Bratsas A, Tousoulis D, Stefanadis C, Manolis AJ, Kallikazaros I. Cardiovascular repercussions of the pseudoexfoliation syndrome. N Am J Med Sci. 2013 Aug;5(8):454-9. doi: 10.4103/1947-2714.117294. PMID 24083219
- [Background] Shazly TA, Farrag AN, Kamel A, Al-Hussaini AK. Prevalence of pseudoexfoliation syndrome and pseudoexfoliation glaucoma in Upper Egypt. BMC Ophthalmol. 2011 Jun 27;11:18. doi: 10.1186/1471-2415-11-18. PMID 21707986
- [Background] Plateroti P, Plateroti AM, Abdolrahimzadeh S, Scuderi G. Pseudoexfoliation Syndrome and Pseudoexfoliation Glaucoma: A Review of the Literature with Updates on Surgical Management. J Ophthalmol. 2015;2015:370371. doi: 10.1155/2015/370371. Epub 2015 Oct 29. PMID 26605078
- [Background] Sangal N, Chen TC. Cataract surgery in pseudoexfoliation syndrome. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):403-8. doi: 10.3109/08820538.2014.959189. PMID 25325866